CLINICAL TRIAL: NCT05198479
Title: A Biomarker Enrichment, Phase II Study of 177Lu-DOTATATE in Metastatic Nasopharyngeal Cancer With a Safety Run-in
Brief Title: Phase II 177Lu-DOTATATE Study in Metastatic NPC With a Safety Run-in
Acronym: SG-AAA-II-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Novartis (Industry); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG-AAA-II-01
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Nasopharyngeal Cancer
Keywords: Peptide Receptor Radionuclide therapy (PRRT); 177Lu-DOTA0-Tyr3-Octreotate; Radionuclide therapy; Metastatic Nasopharyngeal Carcinoma; Theragnostics
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 177 Lu-DOTA0-Tyr3-Octreotate (Experimental): Treatment with 177Lu-DOTATATE consist of a cumulative dose of 23.68 - 29.6 GBq (640 - 800 mCi) 177Lu-DOTA0-Tyr3-Octreotate; Four administrations of 5.92 - 7.4 GBq (160 - 200 mCi) 177Lu-DOTA0-Tyr3-Octreotate; Concomitant amino acids will be given with each administration for kidney protection; 177Lu-DOTA0-Tyr3-Octreotate will be administered at 8±1-week intervals, which can be extended up to 16 weeks to accommodate resolving acute toxicity.
  Interventions: Radiation: 77 Lu-DOTA0-Tyr3-Octreotate

INTERVENTIONS:
Radiation: 77 Lu-DOTA0-Tyr3-Octreotate — Treatment will consist of a cumulative dose of 23.68 - 29.6 GBq (640 - 800 mCi) 177Lu-DOTA0 -Tyr3-Octreotate; Four administrations of 5.92 - 7.4 GBq (160 - 200 mCi) 177Lu-DOTA0-Tyr3-Octreotate; Concomitant amino acids will be given with each administration for kidney protection; 177Lu-DOTA0-Tyr3-Octreotate will be administered at 8±1-week intervals, which can be extended up to 16 weeks to accommodate resolving acute toxicity.

SUMMARY:
This study is the first phase II study of 177Lu-DOTA0-Tyr3-Octreotate in metastatic NPC. Patients whom have failed 2 or more lines of therapy or exhausted standard therapy and are avid on 68Ga-DOTATATE imaging will be eligible to receive up to 4 cycles of 177Lu-DOTA0-Tyr3-Octreotate. The primary outcome will be progression free survival at 6 months.

DETAILED DESCRIPTION:
This would be an open label, single arm, single centre, phase II study designed to evaluate the efficacy of 177Lu-DOTA0-Tyr3-Octreotate in Metastatic NPC.

Patients will first need to go for a 68Ga-DOTATATE scan to determine if they are suitable for 177Lu-DOTA0-Tyr3-Octreotate therapy. A'Hern single stage phase II design (A'Hern, 2001) will be used for conducting the trial. The null hypothesis that the true PFS rate at 6 months is 10% will be tested against the alternate hypothesis of 25%. A total number of 25 patients will be recruited. If there are 5 or more patients who are alive and progression free among these 25 patients at 6 months, we reject the null hypothesis and claim that the treatment is promising.

The design controls the type I error rate at 9.8% and yields a power of 78.6% when the true PFS rate at 6 months is 25%. The first 5 patients will receive 180mCi of 177Lu-DOTA0-Tyr3-Octreotate for the first cycle followed by 200mCi for the remaining 3 cycles if there are no > Grade 2 toxicities after the first cycle. If there are >G2 toxicities, the remaining cycles will proceed at 180mCi. A safety review will be done after the first 5 patients. If there are no significant toxicities, the remaining patients will receive 200mCi for 4 cycles. If there are significant toxicities in patients receiving 200mCi for the 2nd to 4th cycle, the remaining patients will receive 180mCi for 4 cycles. If there are significant toxicities in patients receiving 180mCi for the 2nd to 4th cycle, the remaining patients will receive 160mCi for 4 cycles. Dosimetry scans will be done after each cycle of 177Lu-DOTA0-Tyr3-Octreotate at 1h and 96h. Safety and tolerability of 177LuDOTA0-Tyr3-Octreotate will be assessed for the duration of study treatment.

FDG PET/CT scan and 68Ga-DOTATATE scan will be performed at baseline and after cycle 1 (week 4) and cycle 4 (week 28). CT scans will be done at week 12, 24, then 3-monthly starting from week 40. 177Lu-DOTA0-Tyr3-Octreotate treatment will be continued until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment is permitted. A treatment cycle is eight weeks (56 days) and will be repeated without therapy interruption for 4 cycles unless there is dose limiting toxicities.

ELIGIBILITY:
Inclusion Criteria:

* a histologically confirmed diagnosis of NPC
* metastatic NPC that has failed two or more lines of therapy or exhausted standard therapy
* an Eastern Cooperative Oncology Group performance status of 0-2
* age 21-75 years, a life expectancy of more than 3 months
* no prior use of radionuclide therapy
* no prior radiotherapy to more than 25% of bone marrow
* less than 50% of bone marrow involved on 68Ga-DOTATATE scan
* Krenning score ≥ 3 and at least 75% concordance between 68Ga-DOTATATE scan and 18F-FDG PET scan
* at least 1 bidimensionally measurable (2 cm) site of disease.
* A wash-out period of at least 3 weeks from the last dose of prior chemotherapy is required before the administration of the first dose of 177Lu-DOTATATE.
* adequate hematologic, renal, and liver function using standard laboratory measurements
* no history of other malignancy, except treated basal cell and squamous cell skin carcinomas

Exclusion Criteria:

* Serum creatinine >120 μmol/L or 1.2 mg/dL, or a measured creatinine clearance (or measured glomerular filtration rate (GFR) using plasma clearance methods, not gamma camera-based) of <50 mL/min.
* Hb concentration <5.0 mmol/L (<8.0 g/dL); WBC <3x10^9/L (3000/mm3); platelets <75x10^9/L (75x10^3/mm3).
* Total bilirubin >3 x ULN.
* Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
* Pregnancy (see protocol Appendix 6).
* For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients, who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel) as defined in Appendix 6.
* Peptide receptor radionuclide therapy (PRRT) at any time prior to enrolment in the study.
* Targeted surgery, radiotherapy (external beam), chemotherapy, embolization, interferons, mTOR-inhibitors or other investigational therapy within 3 weeks prior to enrolment in the study.
* Known brain metastases, unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrolment in the study. Patients with a history of brain metastases should have a head CT/MRI to document stable disease prior to enrolment in the study.
* Uncontrolled congestive heart failure (NYHA II, III, IV).
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
* Any patient receiving treatment with short or long acting somatostatin analogs.
* Patients with any other significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
* Urinary incontinence.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
* Patients who have not provided a signed an informed consent form to participate in the study, obtained prior to the start of any protocol related activities.
* Patients who are unable to comply with relevant contact precautions post Lutetium therapy.
* Patients with a synchronous local nasopharyngeal recurrence, with prior high-dose irradiation to the primary tumour.
* Patients with active Hepatitis B (HBsAg positive) or Hepatitis C (HCV Ab positive) infection will be excluded.
* Patients with known history of Human Immunodeficiency Virus (HIV) will be excluded.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS). | Within 76 weeks of start of study treatment.
  PFS is defined as the time from the date of initiating study treatment to the date of documented disease progression as determined by RECIST Criteria, Version 1.1 or death from any cause.
  Point estimates for median PFS and PFS rate at 6 month, with corresponding 95% Confidence Intervals (CIs), will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Objective Response Rate (ORR). | Within 76 weeks of start of study treatment.
  ORR is defined as the percentage of patients who had a partial response or complete response according to RECIST 1.1.
  The ORR and 95% CI will be calculated.
Time to Tumour Progression (TTP) | Within 76 weeks of start of study treatment.
  TTP is defined as the time (number of days) from start of study treatment to objective tumour progression.
Overall Survival (OS). | Within 76 weeks of start of study treatment.
  OS is defined as the time from the date of start of study treatment to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tan, BSc, MBBS, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided